CLINICAL TRIAL: NCT02753660
Title: Comparison Between Pendant Position and Traditional Sitting Position for Successful Spinal Puncture in Spinal Anaesthesia for Cesarean Section
Brief Title: Pendant Position and Traditional Sitting Position for Successful Spinal Puncture in Spinal Anaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Pryambodho Pryambodho, Consultant, Anesthesiologist, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes001
Record Dates: First submitted 2016-04-26; First posted 2016-04-28 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Pregnancy, Caesarean Section
Keywords: spinal, anesthesia, pendant, spinal-bone contact, puncture

ARMS (2):
- Traditional sitting position (Active Comparator): Patient is positioned with her knees flexed 90o, both feet hanging of the bed and propped up by a chair, both arms hugging a pillow, adducted pelvic, maximum pelvic flexion were done to create maximal sagittal lumbal flexion before spinal anesthesia begun.
  Interventions: Procedure: Traditional sitting position
- Pendant position (Experimental): Patients sit with both their underarms propped up on a metal prop, thus both arms hanging from the prop before spinal anesthesia begun.
  Interventions: Procedure: Pendant position

INTERVENTIONS:
Procedure: Traditional sitting position — Subjects were set on traditional sitting position before spinal anesthesia begun.
  Arms: Traditional sitting position
Procedure: Pendant position — Subjects were set on pendant position before spinal anesthesia begun.
  Arms: Pendant position

SUMMARY:
The aim of this study was to compare the successful spinal puncture among patients with pendant position in comparison with those who used traditional sitting position for caesarean section.

DETAILED DESCRIPTION:
Approval from Ethical Committee of Faculty of Medicine University of Indonesia was acquired prior conducting the study. Subjects were given informed consent before enrolling the study. Subjects were divided into Group A for traditional sitting position (n=154) and Group B for pendant position (n=154). The outcome parameters recorded were the number of attempt for the successful spinal puncture, the number of spinal needle-bone contact and the duration to perform spinal puncture. Data were analyzed by using Statistical Package for Social Scientist (SPSS) version 21.0. Numerical data was served in median with minimal and maximal value. Numerical data was analyzed by using Mann-Whitney test. Categorical data was served by using relative risk (RR) with 95% confidence interval (95% CI) and was analyzed by using Chi-Square test.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women aged 18-45 years old
* Body Mass Index (BMI) 18-35 kg/m2
* physical status American Society of Anesthesiologists (ASA) I-III
* planned to undergo cesarean section with spinal anesthesia and signed the informed consent form

Exclusion Criteria:

* Patients with any contraindication for spinal anesthesia (infection on injection site, coagulation disorder, severe hypovolemia, increased intracranial pressure, aortic and/or mitral stenosis)
* pregnancy with head entrapment of the fetus, umbilical cord prolapse, feet presentation,
* Patient with eclampsia
* Patient with cardiovascular diseases
* Patient with scoliosis
* Patient with history of lumbar surgery
* Patient with unpalpable intervertebral space due to thick fatty tissue or edema.

Drop out criteria:

- spinal block was failed or only partial block

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 308 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Successful spinal puncture attempt number | 2 months
  The number of attempt for the successful spinal puncture for each positions
The number of spinal needle-bone contact | 2 months
  The number of spinal needle-bone contact for each positions
Spinal puncture duration | 2 months
  the duration to perform spinal puncture for each positions

CONTACTS AND LOCATIONS:
Overall Officials: Pryambodho Pryambodho, Consultant, Principal Investigator — Indonesia University

REFERENCES:
- [Background] de Filho GR, Gomes HP, da Fonseca MH, Hoffman JC, Pederneiras SG, Garcia JH. Predictors of successful neuraxial block: a prospective study. Eur J Anaesthesiol. 2002 Jun;19(6):447-51. doi: 10.1017/s0265021502000716. PMID 12094920
- [Background] Fisher KS, Arnholt AT, Douglas ME, Vandiver SL, Nguyen DH. A randomized trial of the traditional sitting position versus the hamstring stretch position for labor epidural needle placement. Anesth Analg. 2009 Aug;109(2):532-4. doi: 10.1213/ane.0b013e3181ac6c79. PMID 19608828
- [Background] Soltani Mohammadi S, Hassani M, Marashi SM. Comparing the squatting position and traditional sitting position for ease of spinal needle placement: a randomized clinical trial. Anesth Pain Med. 2014 Apr 5;4(2):e13969. doi: 10.5812/aapm.13969. eCollection 2014 May. PMID 24790901
- [Background] Shabanian G, Saadat M. A position for administration of difficult spinal anesthesia. J Clin Diagn Res. 2014 Mar;8(3):190-1. doi: 10.7860/JCDR/2014/5881.4198. Epub 2014 Mar 15. No abstract available. PMID 24783134
- [Background] Grau T, Leipold RW, Horter J, Conradi R, Martin E, Motsch J. The lumbar epidural space in pregnancy: visualization by ultrasonography. Br J Anaesth. 2001 Jun;86(6):798-804. doi: 10.1093/bja/86.6.798. PMID 11573586
- [Background] Tekeoglu I, Adak B, Bozkurt M, Gurbuzoglu N. Distraction of lumbar vertebrae in gravitational traction. Spine (Phila Pa 1976). 1998 May 1;23(9):1061-3; discussion 1064. doi: 10.1097/00007632-199805010-00019. PMID 9589547
- [Background] Shankar H, Rajput K, Murugiah K. Correlation between spinous process dimensions and ease of spinal anaesthesia. Indian J Anaesth. 2012 May;56(3):250-4. doi: 10.4103/0019-5049.98769. PMID 22923823
- [Background] Brooks RR, Oudekerk C, Olson RL, Daniel C, Vacchiano C, Maye J. The effect of spinal introducer needle use on postoperative back pain. AANA J. 2002 Dec;70(6):449-52. PMID 12526150